CLINICAL TRIAL: NCT01140867
Title: A Korean Open-label, Multi-center, Community-based Trial Assessing the Efficacy and Safety of Zonisamide as Adjunctive Therapy in Patients With Uncontrolled Partial Epilepsy
Brief Title: Open-label, Multi-center Trial of Zonisamide as Adjunctive Therapy in Patients With Uncontrolled Partial Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2090-S082-409
Record Dates: First submitted 2010-05-19; First posted 2010-06-10 (Estimated); Results first posted 2011-09-08 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2011-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Zonisamide

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: zonisamide

INTERVENTIONS:
Drug: zonisamide — zonisamide 100 mg tablet

SUMMARY:
The object of this study is to assess the efficacy and safety of zonisamide as adjunctive therapy in patients with uncontrolled partial epilepsy.

DETAILED DESCRIPTION:
The object of this study is to assess the efficacy and safety of zonisamide as adjunctive therapy in patients with uncontrolled partial epilepsy. Subject takes zonisamide for 16 weeks (4 weeks-titration period, 8 weeks maintenance period). Dose range of zonisamide is 100 ~ 400 mg/day and target dose is 300 mg/day. After 16 weeks, zonisamide efficacy is measured by seizure reduction rate (Each type of seizure: simple partial seizures [SPS], complex partial seizures [CPS], simple partial seizures evolving into generalized tonic-clonic convulsions [SGTC] and total seizure frequency), seizure free rate, responder rate, quality of life in epilepsy (QOLIE-31) and investigator's global evaluation scale. Safety of zonisamide in this study will be estimated by adverse event profile, retention rate and dose of exposure. The duration of this clinical study is 2 years including period of subject enrollment.

ELIGIBILITY:
Inclusion criteria:

1. Epilepsy patient over 15 years old who agrees with Informed Consent Form
2. Patient who has classifiable uncontrolled partial epilepsy according to International Classification of Epileptic Seizures.
3. Patient who has 3 ~ dozens of partial seizure (average more than once seizure per 4 weeks) last 12 weeks despite taking 1 ~ 3 antiepileptic drug(s).
4. Patient who takes 1 ~ 3 marketed antiepileptic drug(s) excluding zonisamide at point of enrollment time.
5. Before study visit, patient who takes stable dose of antiepileptic drug more than 4 weeks.

Exclusion criteria:

1. Patient who has progressive central nervous system (CNS) disorder and/or degenerative disease of the brain.
2. Patient who experiences pseudoseizures and/or who has uncountable clusters.
3. Patient who has serious systemic or drug metabolism affecting disorder .
4. Upward of doubled normal glutamic oxaloacetic transaminase (GOT), glutamic pyruvic transaminase (GPT), bilirubin, blood urea nitrogen (BUN), creatinine levels.
5. Patient who has absolute neutrophil counts <1800/mm3 or platelets <100,000/mm3.
6. Patient who has medical history of renal stones.
7. Patient who is allergic to sulfonamide.
8. Medical history of medicinal poisoning and/or alcoholism and/or serious psychological disorder.
9. Pregnant women, lactating women, women of childbearing age who do not use a preventive method of conception.
10. A terminal patient and/or a scheduled surgical patient.
11. Patient who has medication history of zonisamide.
12. Patient who participated other clinical trial within the last 12 weeks at point of enrollment time of this study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2008-02-29 (Actual); Primary Completion 2010-08-31 (Actual); Study Completion 2011-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jihee Mun, Study Director — Medical Department, Eisai Korea Inc.
Locations (10):
- South Korea (10):
  - Dong-A University Hospital, Dept. of Neurology, Busan
  - Inje Univ. Pusan Paik Hospital, Dept. of Neurology, Busan
  - Keimyung Univ.Dongsan Medical Centre, Dept. of Neurology, Daegu
  - Kyungpook Natl. Univ. Hosp., Dept. of Neurology, Daegu
  - Yeungnam Univ. Medical Center, Dept. of Neurology, Daegu
  - Gachon Medical School Gil Medical Centre, Dept.of Neurology, Incheon
  - Natl. Health Insurance Corporation Ilsan Hosp., Dept. of Neurology, Koyang
  - Bundang CHA Hospital, Dept. of Neurology, Seongnam
  - Kangdong Sacred Heart Hosp., Dept. of Neurology, Seoul
  - Severance Hospital, Dept. of Neurology, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 10 centers in Korea during the period of February 2008 to August 2010.
Groups:
- Zonisamide: Initial dose was 100mg/day, increased by 100mg in week 2 and 4. The target dose was 300mg/day, and the maximum dose was 400mg/day.
Period: Overall Study
Arm/Group | Zonisamide
Started | 121
Completed | 88
Not Completed | 33
Not completed — Adverse Event | 22
Not completed — Lack of Efficacy | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1
Not completed — Uncooperative patient | 2
Not completed — Medication Noncompliance | 2

BASELINE CHARACTERISTICS:
Arm/Group | Zonisamide
Number analyzed (Participants) | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.70 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 121
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Seizure Reduction Rate
Description: The percentage of the seizure reduction after Zonisamide treatment comparing baseline seizure frequency.
Time Frame: Baseline and 16 weeks
Population: Efficacy analyses were based on the FAS (Full analysis set) population, which was comprised of all patients who administrated Zonisamide at least once and reached the maintenance period to evaluate the primary endpoint.
Measure: Mean (Standard Deviation); unit: Percentage of Seizure Reduction Rate
Arm/Group | Zonisamide
Number analyzed (Participants) | 102
Percentage of Seizure Reduction Rate | -16.35 (436)

2. Secondary Outcome: Seizure Free Rate
Description: The percentage of the participants who experienced no seizure during the trial.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Zonisamide
Number analyzed (Participants) | 102
Percentage of Participants | 24.51

3. Secondary Outcome: Responder Rate
Description: The percentage of participants whose median percentage change in seizure frequency after Zonisamide treatment is reduced over 50%.
Time Frame: Baseline and 16 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Zonisamide
Number analyzed (Participants) | 102
Percentage of Participants | 61.76

4. Secondary Outcome: QoL-QOLIE31 (Quality of Life in Epilepsy)
Description: Quality of life assessment tool. Overall scores is calculated by summing subsections, and it ranges from 0 to 100. Higher score presents higher quality of life.
Time Frame: Baseline and 16 weeks
Population: Efficacy analyses were based on the FAS (Full analysis set) population, which was comprised of all patients who administrated Zonisamide at least once and reached the maintenance period to evaluate the primary endpoint. Regarding QOLIE-31, among FAS population, the patients who have both of baseline and 16 week evaluation are included.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Zonisamide
Number analyzed (Participants) | 102
Units on a Scale
  Baseline- Pre-QOLIE 31 total score (N=90) | 56.67 (15.97)
  16 weeks - Post- QOLIE 31 total score (N=90) | 57.70 (15.74)

ADVERSE EVENTS:
Arm/Group | Zonisamide
Serious Adverse Events (participants affected / at risk) | 2/121
Other Adverse Events (participants affected / at risk) | 78/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide (N=121)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (3)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide (N=121)
Dizziness (Nervous system disorders) | 34 (37)
Somnolence (Nervous system disorders) | 29 (32)
Headache (Nervous system disorders) | 17 (23)
Vomiting (Gastrointestinal disorders) | 16 (16)
Anorexia (Metabolism and nutrition disorders) | 22 (25)
Asthenia (General disorders) | 8 (8)
Weight decreased (Investigations) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No